CLINICAL TRIAL: NCT02081703
Title: A Phase 2 Study to Evaluate the Safety & Efficacy of Two Dose/Volume Levels of a Single Intrathecal Preoperative Administration of AYX1 Injection in Patients Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Study to Evaluate Safety/Efficacy of a Single Pre-Op Dose of AYX1 Injection to Treat Pain After Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adynxx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADYX-003
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Postsurgical Pain
Keywords: Postsurgical pain; Total knee arthroplasty; Total knee replacement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AYX1 Injection 660 mg / 6 mL (Experimental): Single Intrathecal (spinal) administration of AYX1 Injection (660 mg in 6 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: AYX1 Injection 660 mg / 6 mL
- Placebo Injection 6 mL (Placebo Comparator): Single Intrathecal (spinal) administration of Placebo Injection (6 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: Placebo Injection 6 mL
- AYX1 Injection 1100 mg / 10 mL (Experimental): Single Intrathecal (spinal) administration of AYX1 Injection (1100 mg in 10 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: AYX1 Injection 1100 mg / 10 mL
- Placebo Injection 10 mL (Placebo Comparator): Single Intrathecal (spinal) administration of Placebo Injection (10 mL) just prior to intrathecal administration of spinal anesthetic for knee surgery
  Interventions: Drug: Placebo Injection 10 mL

INTERVENTIONS:
Drug: AYX1 Injection 660 mg / 6 mL — 6 mL solution for intrathecal injection with 660 mg of AYX1
  Arms: AYX1 Injection 660 mg / 6 mL
Drug: AYX1 Injection 1100 mg / 10 mL — 10 mL solution for intrathecal injection with 1100 mg of AYX1
  Arms: AYX1 Injection 1100 mg / 10 mL
Drug: Placebo Injection 6 mL — 6 mL solution for intrathecal injection; Vehicle formulation designed to mimic AYX1 Injection (with no active drug)
  Arms: Placebo Injection 6 mL
Drug: Placebo Injection 10 mL — 10 mL solution for intrathecal injection; Vehicle formulation designed to mimic AYX1 Injection (with no active drug)
  Arms: Placebo Injection 10 mL

SUMMARY:
The objectives of this study are to evaluate the safety and analgesic efficacy of a single preoperative intrathecal administration of AYX1 Injection at two dose/volume levels.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary unilateral TKA for painful osteoarthritis without congenital knee pathology
* American Society of Anesthesiologists Physical Status Classification System ≤ 3
* Medically stable as determined by the Investigator based on pre-study medical history, physical/neurological examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings
* Body Mass Index of 18-40 kg/m2
* Stable medical regimen for at least 1 month before randomization
* Able to read and understand study instructions in English, and willing and able to comply with all study procedures

Exclusion Criteria:

* More than 2 other current focal areas of pain, none greater in intensity than the target knee and no other active chronic pain conditions that would compromise operative knee pain evaluation
* Inflammatory arthridities (e.g., rheumatoid arthritis, lupus, ankylosing spondylitis, psoriatic arthritis), with the exception of clinically stable/non-active gout that does not affect the knee and does not interfere with walking
* Operative arthroscopy in the surgical knee in the last 4 months (except for meniscal repair which will be no shorter than 6 months before randomization) or in the contralateral knee in the last 2 months (or 3 months for meniscal repair), or other prior surgery in either knee in the last 12 months, except for diagnostic arthroscopy
* Planned use of any of the following for TKA: general anesthesia using potent inhalational agents, peripheral nerve block (i.e., femoral nerve block), neuroaxial (intrathecal or epidural) opioids postoperatively, or knee capsule injections
* Received aspirin or any nonsteroidal anti-inflammatory drug (NSAID) prior to randomization within the washout period required by the surgical team for surgery with spinal anesthetic, or planned use of NSAIDS post-operatively through Day 28
* Use of more than 20 mg per day (on average) of oral morphine or its equivalent within 1 month prior to randomization
* Use of adjuvant analgesics for chronic pain control (e.g., gabapentin, pregabalin) within 2 weeks prior to randomization or planned use post-operatively through Day 28
* Daily use of benzodiazepines in the 3 months prior to randomization (unless used for sleep and dosage will be consistent after surgery)
* Use of systemic corticosteroids (does not include inhaled steroids) within 3 months or intra-articular steroid injections within 1 month prior to randomization, or planned use of either post-operatively through Day 28
* Treatment with immunosuppressives, antipsychotics, anticholinergics, or anticonvulsants within 1 month of randomization, with the exception of aspirin for cardiac prophylaxis (as long as discontinued within 1 week of randomization)
* Current neurologic disorder, which could confound the assessment of pain (e.g., Parkinson's, Multiple Sclerosis)
* Current active depression symptoms
* Has had a change in dose or regimen of SSRIs or SNRIs for depression within 1 month of randomization
* Mini Mental State Exam score < 24 at Screening
* Severe pulmonary disease; if symptomatic sleep apnea is currently treated with continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BIPAP), use must be continued postoperatively at least during the inpatient period. Patients with sleep apnea associated with a history of postoperative delirium are excluded.
* Current evidence of alcohol abuse or history of alcohol-related complications within 1 year of randomization including, but not limited to, alcoholic withdrawal seizures, hallucinations, delirium tremens or detoxification treatment
* Known or suspected history of illicit drug abuse within 1 year before randomization, current or planned use of medical marijuana, or history of opioid dependence within 2 years before randomization
* Any malignancy within the past year, with the exception of basal cell carcinoma or uncomplicated or stable skin cancers documented to not require further or immediate treatment
* Women who are pregnant or nursing
* Previous participation in any study involving AYX1 Injection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain with walking during 5 meter walk test | 0-48 hours after surgery
  Mean pain rating on the Numerical Rating Scale (NRS) with walking during the 5 meter walk test during the inpatient stay (0-48 hours)
Pain with walking during 15 meter walk test | Hospital Discharge to Day 28
  Mean pain rating on the Numerical Rating Scale (NRS) with walking during the 15 meter walk test during the outpatient period up to Day 28

SECONDARY OUTCOMES:
Pain with 45 degrees of knee flexion | 0-48 hours after surgery
  Mean pain rating on the Numerical Rating Scale (NRS) for 45 degrees passive knee flexion during the inpatient stay
Pain with 90 degrees of knee flexion | Hospital discharge to Day 28
  Mean pain rating on the Numerical Rating Scale (NRS) for 90 degrees passive knee flexion during the outpatient period to Day 28
Total use of opioid medications (morphine equivalents) during hospital stay | 0-48 hours after surgery
Total use of opioid medications (morphine equivalents) post-discharge to Day 28 | Hospital Discharge to Day 28

OTHER OUTCOMES:
Percentage of subjects achieving 90 degrees of knee flexion | Hospital discharge to Day 42
  Percentage of subjects achieving 90 degrees of active knee flexion in the operative knee at Discharge through Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Manning, MD, PhD, Study Director — Adynxx, Inc.
Locations (2):
- United States (2):
  - Sheffield, Alabama
  - Phoenix, Arizona